CLINICAL TRIAL: NCT01932216
Title: Cosmesis, Patient Satisfaction and Quality of Life After da Vinci Single Site and Multiport Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISI-RCTSS-001
Record Dates: First submitted 2013-08-27; First posted 2013-08-30 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Symptomatic Gallbladder Disease
Keywords: robotic single-site cholecystectomy; laparoscopic cholecystectomy; cosmesis; quality of life
MeSH Terms: interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-site robotic cholecystectomy (Active Comparator): Single-site cholecystectomy using da Vinci robotic assisted surgery
  Interventions: Procedure: Cholecystectomy
- Multi-port laparoscopic cholecystectomy (Active Comparator): Multi-port cholecystectomy using laparoscopic surgery
  Interventions: Procedure: Cholecystectomy

INTERVENTIONS:
Procedure: Cholecystectomy — Gallbladder removal

SUMMARY:
Prospective, randomized , multicenter study comparing cholecystectomy performed with da Vinci Single Site Instruments™ to multi-port (four ports) laparoscopy

DETAILED DESCRIPTION:
Prospective, randomized , multicenter study comparing cholecystectomy performed with da Vinci Single Site Instruments™ to multi-port (four ports) laparoscopy.

* The primary objective of this study is to evaluate cosmesis, patient satisfaction and quality of life after robotic- assisted single incision cholecystectomy procedure using da Vinci Single- Site Instruments™ in comparison to a multiport laparoscopic approach.
* The secondary objective of this study is to assess the peri-operative clinical outcomes of robotic- assisted single incision cholecystectomy with da Vinci Single - Site Instruments™ in comparison to a multiport laparoscopic approach.
* The third objective of this study is to evaluate hernia incidence at 1 year and 18 months after surgery

ELIGIBILITY:
Inclusion Criteria:

* Patient between ages of 18- 80 year
* Patient with symptomatic gallbladder disease
* Patient willing to participate in this study and able to provide informed consent

Exclusion Criteria:

* Patient pregnancy
* Emergency patient
* Patient with acute cholecystitis
* Patient with upper midline visible abdominal scars or keloid
* Presence of umbilical hernia , or prior umbilical hernia repair
* Inability of patients to tolerate Trendelenberg position or pneumoperitoneum
* Patient with cirrhosis
* Patients with mental impairment that preclude giving informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Cosmesis | up to 3 months after surgery
  The primary objective of this study is to evaluate cosmesis, patient satisfaction and quality of life after robotic- assisted single incision cholecystectomy procedure using da Vinci Single- Site Instruments™ in comparison to a multiport laparoscopic approach.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - Huntington Memorial Hospital, Pasadena, California
  - JFK Medical center, Lake Worth, Florida
  - Baptist Health South Florida, Miami, Florida
  - West Suburban Hospital, Elmwood Park, Illinois
  - Dr. Omar Kudsi, Brockton, Massachusetts
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Drexel University, Philadelphia, Pennsylvania
- Athens Medical center, Marousi, Athens, Greece

REFERENCES:
- [Derived] Kudsi OY, Castellanos A, Kaza S, McCarty J, Dickens E, Martin D, Tiesenga FM, Konstantinidis K, Hirides P, Mehendale S, Gonzalez A. Cosmesis, patient satisfaction, and quality of life after da Vinci Single-Site cholecystectomy and multiport laparoscopic cholecystectomy: short-term results from a prospective, multicenter, randomized, controlled trial. Surg Endosc. 2017 Aug;31(8):3242-3250. doi: 10.1007/s00464-016-5353-4. Epub 2016 Nov 18. PMID 27864724